CLINICAL TRIAL: NCT05847192
Title: Tau Networks in Psychotic Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Jeremy Koppel, Assistant Professor, Northwell Health
Other Study IDs: 22-0394_AFA
Record Dates: First submitted 2023-04-17; First posted 2023-05-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease; Alzheimer Disease With Delusions; Alzheimer Disease With Psychosis
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected and tested for APOE genotype in order to stratify participants by APOE allele status during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Alzheimer's disease: * Age 65-85 years old.
  * Diagnosis of probable AD dementia according to NIA-AA criteria.
  * Mini-Mental State Examination (MMSE) score ≥ 10 and ≤ 26 at the screening visit.
  * Clinical Dementia Rating (CDR) score ≥ 0.5.
  * Logical Memory delay score of ≤8 for 16+ years of education, ≤4 for 8-15 years of education, and ≤2 for 0-7 years of education
  Participants will undergo neuropsychological examination, blood collection, sensorimotor gating/ERP testing, MRI and [18F]-PI2620 PET scan.
  Interventions: Diagnostic Test: [18F]-PI2620 PET scan
- Alzheimer's disease with psychosis: - All the criteria for AD are met.
  Presence of one (or more) of the following symptoms:
  * Visual or auditory hallucinations (e.g., seeing silent individuals standing in the room, seeing children in the yard, or seeing animals in the house).
  * Delusions (fixed false beliefs that the patient believes to be true, e.g., that the spouse is unfaithful, that possessions are being stolen, or that one is not who one claims to be).
  Participants will undergo neuropsychological examination, blood collection, sensorimotor gating/ERP testing, MRI and [18F]-PI2620 PET scan.
  Interventions: Diagnostic Test: [18F]-PI2620 PET scan
- Cognitively Unimpaired Healthy: Age 65-85 years old.
  * No known genetic risk factors for dementia.
  * No cognitive complaint
  * Mini-Mental State Examination (MMSE) score ≥ 26 at the screening visit.
  * Logical Memory delay score of ≥9 for 16+ years of education, ≥5 for 8-15 years of education, and ≥3 for 0-7 years of education
  Participants will undergo neuropsychological examination, blood collection, sensorimotor gating/ERP testing, MRI and [18F]-PI2620 PET scan.
  Interventions: Diagnostic Test: [18F]-PI2620 PET scan

INTERVENTIONS:
Diagnostic Test: [18F]-PI2620 PET scan — The PET scan will measure the regional distribution of tau aggregation in AD patients with and without psychosis compared to Cognitively Unimpaired Healthy participants with the PET radiotracer [18F]-PI2620.

SUMMARY:
This research project aims to understand the brain mechanisms behind the manifestation of psychotic symptoms in Alzheimer´s disease (AD), and nature of the unique relationship with tau pathology. Amongst the cognitive manifestations of psychosis are impairments related to frontal circuits (social cognition, working memory and executive function deficits). The investigator's previous work suggests a role of tau pathology (one of the hallmarks of AD neuropathology) in the manifestation of psychosis in AD. However, the cerebral mechanisms that underly this association remain poorly understood. The overarching aim of the study is is to investigate the mechanisms by which tau network pathology may promote the presentation of psychosis in AD.

DETAILED DESCRIPTION:
The specific aims of this application are:

1. To measure the regional distribution of tau aggregation in AD patients with psychosis (AD+P) compared to AD without psychosis (AD-P) and Cognitively Unimpaired Healthy (CUH) participants with the PET radiotracer [18F]-PI2620;
2. To measure structural and functional brain networks properties in AD+P compared to AD-P patients and CUH participants using MRI;
3. To examine the association of tau pathology with structural/functional network properties; electrophysiologic biomarkers of neurotransmission and neuroplasticity; and psychotic symptoms. The current project will determine whether identification of tau pathology, and associated network connectivity disruptions and sensorimotor gating impairments, may be informing as potential biomarkers for psychosis in AD. As severe adverse events are associated with atypical antipsychotics in AD psychosis, this work will provide insights into whether anti-tau therapies such as monoclonal antibodies to tau, now being investigated in clinical trials, may be effective in the antipsychotic treatment of AD.

ELIGIBILITY:
Inclusion Criteria Alzheimer´s disease (AD) participants:

* Age 65-85 years old.
* Diagnosis of probable AD dementia according to National Institute on Aging-Alzheimer's Association (NIA-AA) criteria.
* Mini-Mental State Examination (MMSE) score ≥ 10 and ≤ 26 at the screening visit.
* Clinical Dementia Rating (CDR) score ≥ 0.5.
* Logical Memory delay score of ≤8 for 16+ years of education, ≤4 for 8-15 years of education, and ≤2 for 0-7 years of education

Exclusion Criteria Alzheimer´s disease (AD) participants:

* Rosen-modified Hachinski Ischemia Score > 4 at the screening visit.
* History of stroke.
* Evidence of a clinically relevant neurological disorder other than probable AD at the screening visit. Participants with insulin dependent type 2 diabetes, a history of CVD, a history of epilepsy, a history of TBI with greater than 15 minutes of loss of consciousness, a movement disorder, autoimmune disease affecting the CNS, or delirium.
* Evidence of a clinically relevant or unstable psychiatric disorder, based on DSM-5 criteria, including schizophrenia or other psychotic disorder, bipolar disorder, delirium, or current/active major depression.
* History of alcoholism or drug dependency/abuse within the last 5 years before screening.
* Presence of metal implants such as pacemakers, ear implants, internal bullet fragments or shrapnel.
* Inability to lie flat for 1 hour approximately.
* hearing impairment as evidenced by the inability to hear 500, 1000 and 6000 Hz bilaterally on an OAE evaluation. Subjects with hearing aides will be allowed to participate if they meet minimum hearing requirements.

Specific Inclusion Criteria for Alzheimer´s disease (AD) with Psychotic symptoms:

* All the criteria for AD are met.
* Presence of one (or more) of the following symptoms:

  * Visual or auditory hallucinations (e.g., seeing silent individuals standing in the room, seeing children in the yard, or seeing animals in the house).
  * Delusions (fixed false beliefs that the patient believes to be true, e.g., that the spouse is unfaithful, that possessions are being stolen, or that one is not who one claims to be).

Inclusion Criteria Cognitively Unimpaired Healthy (CUH) participants:

* Age 65-85 years old.
* No known genetic risk factors for dementia.
* No cognitive complaint
* Mini-Mental State Examination (MMSE) score ≥ 26 at the screening visit.
* Logical Memory delay score of ≥9 for 16+ years of education, ≥5 for 8-15 years of education, and ≥3 for 0-7 years of education

Exclusion Criteria Cognitively Unimpaired Healthy (CUH) participants:

- Same criteria as AD participants above.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Alzheimer´s disease (AD) participants Alzheimer´s disease (AD) with psychotic symptoms Cognitively Unimpaired Healthy (CUH) participants
Sampling Method: Non-Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Tau PET scan | 5 years
  To measure the distribution of tau aggregation in AD patients with and without psychosis, compared to cognitively unimpaired healthy subjects with the PET radiotracer [18F]-PI2620.

SECONDARY OUTCOMES:
MRI of the brain | 5 years
  To measure brain networks in AD patients with and without psychosis compared to Cognitively Unimpaired Healthy subjects.

OTHER OUTCOMES:
PPI (pre-pulse inhibition) testing | 5 years
  To examine the association of tau pathology with electrophysiologic biomarkers of neurotransmission and neuroplasticity; and psychotic symptoms. The project will determine whether sensorimotor gating impairments may be informative as a potential biomarker for psychosis in AD.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Koppel, MD, Principal Investigator — Northwell Health
Locations (1):
- The Feinstein Institutes for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No